CLINICAL TRIAL: NCT01740154
Title: Exploration of the Neuromuscular Mechanisms Associated With Sunitinib Related Fatigue
Brief Title: Sunitinib Malate Related Fatigue in Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8811; NCI-2012-00988 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Fatigue; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Fatigue; Carcinoma, Renal Cell | interventions — Transcranial Magnetic Stimulation; Neurofeedback; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (sunitinib malate, neuromuscular testing) (Experimental): Patients receive sunitinib malate PO daily for 4 weeks. Patients undergo neuromuscular testing at baseline and on day 28 and complete fatigue assessment at baseline and on days 14 and 28.
  Interventions: Procedure: transcranial magnetic stimulation; Procedure: electromyography; Other: survey administration; Drug: sunitinib malate

INTERVENTIONS:
Procedure: transcranial magnetic stimulation — Undergo TMS
  Other Names: TMS
Procedure: electromyography — Undergo EMG
  Other Names: EMG
Other: survey administration — Ancillary studies
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
The purpose of this research study is to determine how sunitinib (sunitinib malate) causes fatigue. Patients will be asked to complete a brief questionnaire (survey) to rate their levels of fatigue every two weeks while they are participating in this research study. The questionnaire takes approximately 10-15 minutes to complete and is 9 questions. A series of physical measurements for fatigue will be performed before the first dose of sunitinib and again (4) weeks later to see if there are any changes in physical level of fatigues

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the mechanisms associated with sunitinib related fatigue by recording EMG signals during a submaximal elbow contraction, twitch force and TMS prior to and at the end of 4 weeks of sunitinib in metastatic RCC patients.

OUTLINE:

Patients receive sunitinib malate orally (PO) daily for 4 weeks. Patients undergo neuromuscular testing at baseline and on day 28 and complete fatigue assessment at baseline and on days 14 and 28.

.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell cancer with metastases; pathology from either primary or metastatic tumor; no histologic subtype restriction
* Evidence of measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 or evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance score 0 to 1
* Hemoglobin >= 9 gram/dL
* Common Terminology Criteria for Adverse Events (CTCAE) fatigue levels pre-treatment < 2
* Signed and dated informed consent

Exclusion Criteria:

* Greater than 2 previous systemic treatments for RCC
* Heart failure, New York Heart Association (NYHA) class 3 and 4
* Unstable angina (defined as ongoing use of nitrates or cardiac ischemia in the prior 6 months)
* Arrhythmia uncontrolled by medication
* Hypertension (> 160/90 mmHg) not controlled with medical management
* Brain metastases or previous cranial radiation, leptomeningeal cancer
* Surgery within 2 weeks of study entrance
* History of stroke, myasthenia gravis, multiple sclerosis, polyneuropathy
* Pregnancy or breast feeding
* Central-nervous system active medications, intake or withdrawal of which lowers seizure threshold (determination made in consultation with study's responsible treating physician)
* Any history of epilepsy, convulsion or seizure
* Medication-resistant epilepsy in a first-degree relative
* Cochlear implants or internal pulse generators or cardiac pacemakers or intracardiac lines
* Metallic implants in the vicinity of discharging coil in the head or cervical spine
* Unexplained fainting spells/syncope or multiple concussions
* History of severe head trauma (followed by loss of consciousness)
* Implanted brain or spinal cord electrodes/stimulation
* Medication infusion device
* Frequent/severe headaches or severe migraines
* Past or current medical history of diagnosed or undiagnosed tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
Started | 13
Completed | 12
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Patients accrued on study
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants]
  40-49 years | 1
  50-59 years | 5
  60-69 years | 5
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Changes of Muscular (Peripheral) Fatigue Maximal Twitch Force (MTF)
Description: The MTF will be elicited by supramaximal-intensity electrical stimulation of the muscle before and after the sustained contraction (SC). If the muscle is fatigued at the end of the SC, the MTF will be reduced because the ability of muscle to generate force declines with fatigue. If the sunitinib treatment results in minimal muscular fatigue, the MTF will not have as much reduction in the 2nd as that in the 1st session.
Time Frame: Baseline and 28 days
Population: Data not collected
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
Number analyzed (Participants) | 0

2. Primary Outcome: Change in EMG Amplitude and Power Frequency
Description: EMG amplitude will increase (for low-intensity SC) and mean power frequency (MPF) decrease with muscle fatigue. The EMG signals recorded during the SC, its amplitude and MPF will be analyzed to determine their changes at the end vs. beginning of the SC. If the sunitinib results in minimal muscular fatigue, the amount of EMG increase and MPF decrease will be reduced in the 2nd compared with those the 1st session.
Time Frame: Baseline and 28 days
Population: Data not collected
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in Motor Evoked Potential (MEP) by TMS
Description: TMS illustrates the changes in corticospinal excitability occurring in association with fatigue. Central muscle evoked response (MEP) will be elicited using transcranial magnetic stimulation (TMS) using single stimulus pulses applied to the scalp overlying the primary motor cortex.
Time Frame: Baseline and 28 days
Population: Data not collected
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Supportive Care (Sunitinib Malate, Neuromuscular Testing)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Sunitinib Malate, Neuromuscular Testing) (N=13)
Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Sunitinib Malate, Neuromuscular Testing) (N=13)
Fatigue (General disorders) | 12 (16)

LIMITATIONS AND CAVEATS:
Data not collected for outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes